CLINICAL TRIAL: NCT06701552
Title: MIH Prevalence Among Early Adulthood Patients Attending Cairo University Dental Educational Hospital and Its Correlation to Dental Caries Experience: a Cross-Sectional Study
Brief Title: Prevalence of MIH in Young Adults At Cairo University Dental Hospital and Its Link to Dental Cavities: a Cross-Sectional Study
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Norhan zaki helmy zaki, dentist, Cairo University
Other Study IDs: 14422018483276
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Molar Incisor Hypomineralization; Dental Caries
Keywords: MIH
MeSH Terms: conditions — Molar Hypomineralization; Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — There is no sample to be retained as this is a cross sectional study aiming to know the prevalence of MIH among young adults and its correlation to caries prevalence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- A Group of 266 young adult Egyptian patients: Patients will be examined for prevalence of molar incisor hypomineraliztion and its correlation to caries incidence

SUMMARY:
We are conducting a study to understand how often MIH (Molar Incisor Hypomineralization) occurs and whether it is linked to a higher chance of dental cavities (caries).

MIH is a condition where the enamel (the hard outer surface) of the first permanent molars and incisors (front teeth) doesn't develop properly, making these teeth more prone to damage and decay. We are looking at whether patients with MIH have more cavities in their teeth compared to patients without MIH.

This study aims to help us learn more about the connection between MIH and dental health, so we can improve care and prevention strategies for kids at risk of cavities.

ELIGIBILITY:
Inclusion Criteria:

* patients whose age between 18 and 30 years old provide informed consent Egyptian patients from both sexes

Exclusion Criteria:

* patients under or over this age group patients undergoing orthodontic treatment patients who refuse to participate

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Egyptian participants whose between 18 and 30 years old, both sexes will be included
Sampling Method: Probability Sample
Enrollment: 266 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
prevalence of MIH | one year
  Prevalence of MIH among patients will be described as a percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes